CLINICAL TRIAL: NCT00973245
Title: BAY 59-7939 (Factor Xa Inhibitor) Phase II Once Daily Dose Study in Patients With Atrial Fibrillation
Brief Title: BAY59-7939 in Atrial Fibrillation Once Daily (OD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11866
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation
Keywords: BAY59-7939; Rivaroxaban; Non-valvular atrial fibrillation; Japanese Patients; Phase II
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)
- Arm 2 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)
- Arm 4 (Active Comparator)
  Interventions: Drug: Warfarin
- Arm 3 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)

INTERVENTIONS:
Drug: Xarelto (Rivaroxaban, BAY59-7939) — 10mg od
  Arms: Arm 1
Drug: Xarelto (Rivaroxaban, BAY59-7939) — 15mg od
  Arms: Arm 2
Drug: Xarelto (Rivaroxaban, BAY59-7939) — 20mg od
  Arms: Arm 3
Drug: Warfarin — Dose-adjusted warfarin based on target INR values
  Arms: Arm 4

SUMMARY:
This is an exploratory investigation of safety, pharmacokinetic (PK) and pharmacodynamic (PD) effects of BAY59-7939 with multiple oral doses of 10 mg, 15 mg and 20 mg once daily (od) in Japanese subjects with non-valvular atrial fibrillation (originally described in Japanese).

ELIGIBILITY:
Inclusion Criteria:

Japanese subjects with non-valvular AF who met all of the following criteria:

* Male subjects aged 20 years or older and postmenopausal female subjects
* Subjects with persistent or paroxysmal non-valvular AF with >/=2 episodes before enrollment, at least 1 of which had been verified by ECG recording within 4 weeks before randomization
* Subjects who were at risk for stroke as follows:
* Subjects with at least one risk factor for thromboembolism (hypertension, diabetes mellitus, coronary artery disease, congestive heart failure).
* Subjects aged 60 years old and above regardless of the existence of above risk factors.

Exclusion Criteria:

* History or presence of stroke or transient ischemic attack.
* History of intracerebral hemorrhage.
* History or presence of bleeding at randomization; intraocular or gastrointestinal bleeding within the last 6 months prior to randomization.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2006-07; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
(Safety) Incidence of bleeding | Throughout treatment and followup period
(PK/PD) BAY 59-7939 concentrations / Factor Xa activity, PT, PT-INR, PTT and HEPTEST | Day 14 and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- Japan (10):
  - Chikushino-shi, Fukuoka
  - Fukuoka, Fukuoka
  - Nōgata, Fukuoka
  - Asahikawa, Hokkaido
  - Kobe, Hyōgo
  - Takarazuka, Hyōgo
  - Kuwana, Mie-ken
  - Sendai, Miyagi
  - Tokorozawa, Saitama
  - Shinagawa-ku, Tokyo